CLINICAL TRIAL: NCT05454735
Title: Perioperative Blood Glucose Variability and Autonomic Nervous System Activity in On-pump Cardiac Surgery Patients: Study Protocol of a Single-center Observational Study.
Brief Title: Glycemic Variability and Autonomic Nervous System in Cardiac Surgery Patients
Acronym: CAESAR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/616
Record Dates: First submitted 2022-06-10; First posted 2022-07-12 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-01

CONDITIONS: Blood Glucose Variability; Cardiac Surgical Procedures; Autonomic Nervous System
MeSH Terms: interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urinary and blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1: patients with known insulin-requiring type 2 diabetes mellitus undergoing planned on-pump coronary artery bypass graft surgery
  Interventions: Procedure: coronary artery bypass surgery
- Group 2: patients with known non-insulin-requiring type 2 diabetes mellitus undergoing planned on-pump coronary artery bypass surgery
  Interventions: Procedure: coronary artery bypass surgery
- Group 3: non-diabetic patients undergoing planned aortic valve replacement surgery
  Interventions: Procedure: aortic valve replacement surgery
- Group 4: non-diabetic patients undergoing planned on-pump coronary artery bypass graft surgery
  Interventions: Procedure: coronary artery bypass surgery

INTERVENTIONS:
Procedure: coronary artery bypass surgery — coronary artery bypass surgery
  Groups: Group 1; Group 2; Group 4
Procedure: aortic valve replacement surgery — aortic valve replacement surgery
  Groups: Group 3

SUMMARY:
On-pump coronary artery bypass graft (CABG) and valve replacement surgeries are high-risk procedures. Among the risk factors for postoperative complications, perioperative hyperglycemia and blood glucose variability have been reported to be associated with increased morbidity and mortality. The treatment of hyperglycemia using intravenous insulin infusion improves the prognosis in cardiac surgery patients. However, the determinants of postoperative blood glucose variability and the mechanisms leading to its deleterious impact are unknown. Thus, to date, there is no therapeutic intervention that could effectively prevent and treat the deleterious impact of glycemic variability on postoperative outcome. The purpose of the study is to evaluate whether perioperative alteration of the autonomic nervous system and preoperative blood glucose variability could be related to perioperative glycemic variability.

DETAILED DESCRIPTION:
The main objective is to describe the relationship between preoperative glycemic variability and glycemic variability during the first 48 postoperative hours.

The secondary objectives are :

1. to describe the relationship between preoperative glycemic variability and glycemic variability during the first 48 hours postoperative according to:

   * diabetic and non-diabetic status
   * the type of surgical intervention
2. to describe the relationship between the parameters evaluating the preoperative activity of the autonomic nervous system and:

   * preoperative glycemic variability
   * glycemic variability during the first 48 postoperative hours
3. to describe the relationship between glycemic variability during the first 48 postoperative hours and:

   * parameters evaluating the activity of the autonomic nervous system during the first 48 postoperative hours
   * diabetes phenotype
   * markers of inflammation
   * markers of endothelial dysfunction
4. to describe the morbidity and mortality within 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planned cardiac surgery
* Age ≥ 18 years old and < 80 years old
* Group 1: patients with known insulin-requiring type 2 diabetes mellitus undergoing planned on-pump coronary artery bypass surgery
* Group 2: patients with known non-insulin-requiring type 2 diabetes mellitus undergoing planned on-pump coronary artery bypass surgery
* Group 3: non-diabetic patients undergoing planned aortic valve replacement surgery
* Group 4: non-diabetic patients undergoing planned on-pump coronary artery bypass surgery

Exclusion Criteria:

* Emergent surgery (less than 48 hours between anesthestetic consultation and surgery)
* Combined surgery (coronary artery bypass graft associated with valve surgery, multiple valve replacement, surgery of the ascending aorta)
* Extreme weight: body mass index (BMI) > 35 kg.m-2 or < 18 kg.m-2.
* Off-pump coronary artery bypass graft surgery
* Type 1 diabetes mellitus
* Patient unable to consent
* Pregnant and/or breastfeeding woman
* Permanent preoperative chronic heart rhythm disorder
* Pacemaker
* Unstable patient condition in preoperative period
* Expected life expectancy less than 48 hours.
* Subject unlikely to cooperate in the study and/or low cooperation anticipated by the investigator.
* Duration of continuous preoperative glycemic recording of less than 48 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic and non-diabetic adult patients undergoing planned on-pump cardiac surgery
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Glycemic variability, measured by subcutaneous blood glucose continuous monitoring sensor, calculated by the coefficient of glycemic variability | From 14 days before surgery (at least 48 hours before surgery) to 7 days after surgery
  Continuous blood glucose monitoring using a subcutaneous blood glucose continuous monitoring sensor (FreeStyle Libre Pro)

SECONDARY OUTCOMES:
Autonomic nervous system activity, measured by non-invasive continuous heart rate monitoring, calculated by measuring the R-R interval | From the day before surgery (at admission in the cardiac surgery department the day before surgery) to Day 3 after surgery
  Continuous non-invasive continuous heart rate monitoring using the MooKy HR memory device will allow the continuous measurement of the R-R interval and the R-R interval variability to quantify the activity of the autonomic nervous system.
Vasopressine blood level | The day before surgery, at admission in the postoperative intensive care unit, at day 1 and at day 2 after surgery
  Vasopressine blood level will be measured from blood samples to assess the relationship between blood glucose variability and endothelial dysfunction.
Autonomic nervous system activity | The day before surgery.
  Compass 31 scale: the Compass 31 scale is a validated clinical scale that allows to identify the degree au autonomic nervous system dysfunction.
Endocan blood level | The day before surgery, and at admission in the postoperative intensive care unit, and at day 1 and at day 2 after surgery.
  Endocan blood level will be measured from blood samples to assess the relationship between blood glucose variability and endothelial dysfunction.
8-iso PGF2a urinary level | The day before surgery, and at admission in the postoperative intensive care unit, and at day 1 and at day 2 after surgery.
  8-iso PGF2a urinary level will be measured from urinary samples to assess the relationship between blood glucose variability and oxidative stress.
IL-6 blood level | The day before surgery, and at admission in the postoperative intensive care unit, and at day 1 and at day 2 after surgery.
  IL-6 blood level will be measured from blood samples to assess the relationship between blood glucose variability and systemic inflammation.
IL-10 blood level | The day before surgery, and at admission in the postoperative intensive care unit, and at day 1 and at day 2 after surgery.
  IL-10 blood level will be measured from blood samples to assess the relationship between blood glucose variability and systemic inflammation.
TNF-alpha blood level | The day before surgery, and at admission in the postoperative intensive care unit, and at day 1 and at day 2 after surgery.
  TNF-alpha blood level will be measured from blood samples to assess the relationship between blood glucose variability and systemic inflammation.
Angiotensine blood level | The day before surgery, and at admission in the postoperative intensive care unit, and at day 1 and at day 2 after surgery.
  Angiotensine blood level will be measured from blood samples to assess the relationship between blood glucose variability and endothelial dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BESCH, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (1):
- Post operative intensive care unit of the cardiac surgery department, Besançon, France